CLINICAL TRIAL: NCT05956925
Title: MOBILE Intervention in College Students With Elevated Blood Pressure: A Pilot Study
Brief Title: MOBILE Intervention in College Students With Elevated Blood Pressure
Acronym: MOBILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1565271
Record Dates: First submitted 2023-06-22; First posted 2023-07-24 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: mhealth; hypertension; college students; self-monitoring; lifestyle modifications
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Intervention group vs control group
Masking Description: No masking was done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Following the educational session, the control group participants' BP, ASA24® Dietary Assessment Tool (ASA24; sodium intake), and pre-test knowledge on HTN will be obtained (using Qualitrics). Four weeks later, the participants were scheduled for a follow-up meeting to collect each participant's BP, ASA24, and post-test knowledge on HTN (using Qualitrics).
- MOBILE Intervention Group (Experimental): Intervention participants were required to take daily BP, provide their motivation level, and send them to the research assistant to receive the appropriate text messages.
  Interventions: Behavioral: Intervention group was asked to take their BP daily and rate their motivation level and communicate with the research assistant. Their level will trigger the appropriate behavioral change SMS prompt.

INTERVENTIONS:
Behavioral: Intervention group was asked to take their BP daily and rate their motivation level and communicate with the research assistant. Their level will trigger the appropriate behavioral change SMS prompt. — The investigators showed participants how to use the Health Mate app, upload Withings BP cuff readings, upload historical data to the cloud, read trend lines in their record, rank their daily motivational level, and answer a brief short message service (SMS) question about whether the participants completed the behavioral change task encouraged by the daily message. A one-page instruction sheet with the research team's contact information was provided. Participants were instructed to take their BP daily, before their first meal and encouraged to avoid prior alcohol and caffeine intake as well as physical activity. The participants were instructed to rate their motivational level as low, moderate, or high via SMS when transmitting their BP value. Their level will trigger the appropriate behavioral change SMS prompt.
  Arms: MOBILE Intervention Group

SUMMARY:
The investigators' long-term goal is to develop tailored interventions to influence self-management behaviors in young adults with elevated blood pressure (BP). The investigators seek to test an intervention, mobile health (mHealth) to Optimize BP Improvement (MOBILE), that takes advantage of existing applications and our prior work to allow participants to (1) perform self-measured BP monitoring; (2) receive feedback from a cloud-based cardiovascular disease (CVD) detection platform; and (3) receive tailored text messages that encourage engagement in BP reduction behavior. mHealth technology provides an ideal way to deliver healthcare interventions to young adults. Text messaging is especially appealing to college students, more than 91% of whom use smartphones as their main communication device. For this study, the investigators will recruit 42 college students, ages 18 to 29, with elevated BP to participate in formative developmental project and then a 4-week two-armed trial of MOBILE. The aims of this study are:

Aim 1. To refine the MOBILE intervention during a formative phase involving 8-10 students. Outcomes will include finalized motivation-level-tailored text messages designed to prompt behavior change and a self-administered motivational scale to be employed in the Aim 2 and Exploratory Aim study.

Aim 2. To evaluate the feasibility of implementing the MOBILE intervention in 32 college students with elevated BP. The investigators will operationalize MOBILE feasibility as: (a) acceptability to participants, (b) participation rate, (c) texts delivered and opened, (d) fidelity to daily BP measurement protocol, (e) reported technical problems and challenges, and (f) recruitment and attrition rates.

Exploratory Aim. To examine the preliminary impact of the MOBILE intervention on BP reduction (primary outcome) along with sodium intake and hypertension (HTN) knowledge improvement (secondary outcomes) among 32 college students with elevated BP. Hypothesis: The intervention group will have a significantly greater reduction in BP and sodium intake and greater increase in HTN knowledge from baseline to completion, compared to control group.

DETAILED DESCRIPTION:
The investigators seek to test an intervention, mHealth to Optimize BP Improvement (MOBILE), that takes advantage of existing applications and our prior work to allow participants to (1) perform self-measured BP monitoring; (2) receive feedback from a cloud-based CVD detection platform; and (3) receive tailored text messages that encourage engagement in BP reduction behavior. mHealth technology provides an ideal way to deliver healthcare interventions to young adults.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 Formative Phase:

* Full-time (≥ 12 credits for undergraduate and ≥ 9 credits for graduate) college student at the University of Nevada, Las Vegas (UNLV)
* Aged 18-29 years.

Aim 2 Inclusion criteria:

* Full-time (≥ 12 credits for undergraduate and ≥ 9 credits for graduate) college student at UNLV
* Aged 18-29 years
* Regular access to a mobile smart-phone with unlimited texting
* Elevated BP (SBP 120-129 mm Hg and diastolic blood pressure [DBP] <80 mm Hg) or undiagnosed HTN stage 1 (SBP 130-139 mm Hg or DBP 80-89 mm Hg). Interested participants who have HTN stage 2 (SBP >140 mm Hg or DBP >90 mm Hg) will need clearance from their primary healthcare provider to participate in the study.

Exclusion Criteria:

Aim 2 Exclusion criteria:

* Taking antihypertensive medication (e.g. angiotensin-converting enzyme [ACE] inhibitors, angiotensin II receptor blockers [ARBs], calcium channel blockers [CCBs], beta-blockers, diuretics, or vasodilators)
* Currently pregnant, lactating, or planning to become pregnant during the study duration
* Having diabetes mellitus, hyperlipidemia, or a life-threatening illness or condition associated with HTN.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieu-My T Tran, PhD, RN, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
The pilot study has limited data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had HTN stage II (SBP >140 mm Hg or DBP >90 mm Hg) during screening and enrollment, but did not provide a health care provider note were not assigned to a group.
Period: Overall Study
Arm/Group | Control | MOBILE Intervention Group
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | MOBILE Intervention Group | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean | 21.7 (2.40) | 24.1 (3.03) | 22.9 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 8 | 14
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 125.5 (12.04) | 131.2 (11.30) | 128.45 (11.81)
  Diastolic Blood Pressure | 80.9 (9.01) | 80.6 (8.70) | 80.7 (8.69)
Hypertension Knowledge-Level Scale (HK-LS) [Mean (Standard Deviation); unit: units on a scale] — Assess all participants' knowledge of hypertension using the Hypertension Knowledge-Level Scale (HK-LS). 6 sub-dimensions: definition, medical treatment, drug compliance, lifestyle, diet, and complications 22-item; Responses; Score ranges from 0-22; Higher scores reflect greater knowledge of HTN.
  Reliability: Cronbach's alpha 0.82 & Validity: good content, face, and construct validity, test re-test reliability (0.79), and discriminative validity (0.27->0.40).
  units on a scale | 17.14 (2.48) | 17.87 (3.07) | 17.52 (2.77)
Daily Sodium Intake [Mean (Standard Deviation); unit: mg] — Using the ASA-24 Dietary Assessment Tool to examine daily sodium intake.
  mg | 3765.5 (1953.08) | 3955.4 (2530.53) | 3863.77 (2232.07)
Body mass index category [Count of Participants; unit: Participants] — Height and weight were collected to calculate participants' BMI.
  Participants
    Underweight | 1 | 0 | 1
    Normal or Healthy Weight | 3 | 4 | 7
    Overweight | 4 | 7 | 11
    Obese | 6 | 4 | 10
Education [Count of Participants; unit: Participants]
  Undergraduate | 14 | 6 | 20
  Graduate | 0 | 9 | 9
Martial Status [Count of Participants; unit: Participants]
  Single | 12 | 11 | 23
  Married or living together | 2 | 3 | 5
  Divorced/Separated | 0 | 1 | 1
Insurance coverage [Count of Participants; unit: Participants] | 12 | 12 | 24
Family History of Heart Disease [Count of Participants; unit: Participants] | 8 | 4 | 12
Daily Caloric Intake [Mean (Standard Deviation); unit: calories] — Using the ASA-24 Dietary Assessment tool to evaluate participants' daily caloric intake.
  calories | 1874.2 (752.16) | 2446.5 (1425.86) | 2160.38 (1155.95)

OUTCOME MEASURES:

1. Primary Outcome: BP Level
Description: BP level (systolic and diastolic BP) was taken using the Withings Wireless BP cuff by the participant in the intervention group.
Time Frame: Average value from 28 days
Population: College students between ages 18-29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control | MOBILE Intervention Group
Number analyzed (Participants) | 14 | 15
mm Hg
  Systolic Blood Pressure | 124.0 (12.31) | 118.7 (11.32)
  Diastolic Blood Pressure | 77.9 (7.90) | 73.7 (7.60)

2. Secondary Outcome: Sodium Intake
Description: ASA24 dietary intake were measured in all participants and sodium intake was evaluated using this measurement.
Time Frame: Average of Day 1 and Day 28
Population: College students between the ages of 18-29.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control | MOBILE Intervention Group
Number analyzed (Participants) | 14 | 15
mg | 3046.2 (1095.85) | 3799.39 (2540.8)

3. Secondary Outcome: HTN Knowledge
Description: Assess all participants' knowledge on HTN using the Hypertension Knowledge-Level Scale (HK-LS). 6 sub-dimensions: definition, medical treatment, drug compliance, lifestyle, diet, and complications 22-item; Responses; Score ranges from 0-22; Higher scores reflect greater knowledge of HTN.
  Reliability: Cronbach's alpha 0.82 & Validity: good content, face, and construct validity, test re-test reliability (0.79), and discriminative validity (0.27->0.40).
Time Frame: Average of Day 1 and Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOBILE Intervention Group
Number analyzed (Participants) | 14 | 15
units on a scale | 19.1 (1.54) | 19.3 (1.35)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Control | MOBILE Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05956925/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05956925/SAP_001.pdf
  • Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05956925/ICF_002.pdf